CLINICAL TRIAL: NCT00472225
Title: Open-Labelled, Multicenter Phase II Study of Rituximab in Patients With Steroid-Refractory Chronic Graft-Versus-Host Disease
Brief Title: Study of Rituximab in Patients With Steroid-Refractory Chronic Graft-Versus-Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Korean Society of Hematopoietic Stem Cell Transplantation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Jong Ho Won M.D., Ph.D., The Korean Society of Hematopoietic Stem Cell Transplantation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHSCT-01-2007
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Steroid-Refractory Chronic GVHD
Keywords: Chronic graft-versus-host disease; rituximab
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Rituximab treatment arm
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab Induction: Rituximab 375 mg/m2 weekly IV for 4 consecutive weeks
  Rituximab Maintenance: Rituximab 375 mg/m2 monthly IV for 4 consecutive months
  Other Names: Mabthera

SUMMARY:
Chronic GVHD is the most common late complication following allogeneic stem cell transplantation. It has features resembling autoimmune disorders such as scleroderma, primary biliary cirrhosis, bronchiolitis obliterans, chronic immunodeficiency etc. Thus, chronic GVHD can lead to debilitating complications such as joint contractures, blindness, end-stage lung disease, etc so that chronic GVHD has a major impact both on survival as well as quality of life. Although its pathogenesis is still poorly unclear, it has been reported since 2000 that B cell-mediated immunity may also contribute to development of chronic GVHD other than T cells. Thus, targeting against B cell may be a useful treatment strategy in the treatment of chronic GVHD.

The purpose of this study is to determine whether rituximab, an anti-CD20 monoclonal kimeric antibody is effective in the treatment of chronic graft-versus-host disease (chronic GVHD) refractory to steroid.

DETAILED DESCRIPTION:
1. STUDY OBJECTIVES

   * Primary Endpoints: To assess the response rate
   * Secondary End points

     * To evaluate the discontinuation of corticosteroid
     * To assess the quality of life
2. Treatment schedule

   * The BSA on the date of every treatment cycle may be used as the same value of baseline BSA, if change of body weight is within 10% of baseline body weight.
   * Treatment schedule consists of induction and maintenance therapy as follows

     * Induction - Rituximab 375 mg/m2 weekly IV for 4 consecutive weeks
     * Maintenance - Rituximab 375 mg/m2 monthly IV for 4 consecutive months

ELIGIBILITY:
Inclusion Criteria:

* All recipients underwent allogeneic stem cell transplantation for haematologic disorders
* All recipients diagnosed as chronic GVHD according to diagnostic criteria proposed by National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic GVHD

  * The presence of one diagnostic sign Or
  * The presence of one distinctive sign (Appendix 1B) with laboratory or histopathologic confirmation in the same or other organ if diagnostic feature is not present
* All patients with chronic GVHD have at least moderate score based on the global scoring system of chronic GVHD
* Recipients refractory or resistant to therapy with corticosteroid

  * Patients had chronic GVHD with the same severity during the last one month while they had received the equivalent of prednisone ≥0.5mg/kg per day or 1mg/kg every other day at least for 30 days or longer
* Informed consent
* Other concomitant medication

  * Patients treated with other immunosuppressive agents (cyclosporine, thalidomide etc) as a combination therapy with corticosteroid must be receiving a dosage that has been stable for at least 1 month prior to screening.

Exclusion Criteria:

* Recipients received donor lymphocyte infusions in the preceding 100 days
* Serious comorbid diseases
* Life expectancy of less than 1 month
* Age < 2 years and > 75 years
* Pregnant or intended to become pregnant
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Ages: 3 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) : Resolution of all signs and symptoms of chronic GVHD Partial response (PR) : Improvement (at least 1 clinical score reduction) in 1 or more organs of involvement and no evidence of worsening in any organ | Response evaluation will be perfomed every 4 weeks during the maintenance of rituximab (the 12th, 16th, 20th, 24st, 36th and 52th week).

SECONDARY OUTCOMES:
Steroid tapering | Within one year after start the first dose of rituximab
Quality of life | Baseline, the 8th and 52th week.
Toxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Won, MD, Principal Investigator — Soon Chun Hyang Hospital, Seoul, Korea
Locations (9):
- South Korea (9):
  - Kyungpook University Hospital, Daegu, Kyungsang-do
  - Busan Baik Hospital, Busan
  - Busan National University Hospital, Busan
  - Chun Nam National University Hospital, Gwangju
  - Samsung Medical Center, Seoul
  - Seoul National University, Seoul
  - Soon Chun Hyang Hospital, Seoul
  - The Catholic University of Korea, Seoul
  - Yonsei University Hospital, Seoul

REFERENCES:
- See also: Home page of the Korean society of hematopoietic stem cell transplantation — http://www.bmt.or.kr